CLINICAL TRIAL: NCT02945293
Title: Cognitive, Behavioral and Aging Effects of Pain Medication in Alcohol Users
Acronym: CAAP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Principal Investigator, Monique Cherrier, Associate Professor, School of Medicine: Psychiatry And Behavioral Sciences, University of Washington
Other Study IDs: STUDY00001018; 5R01AG047979 (NIH)
Record Dates: First submitted 2016-10-18; First posted 2016-10-26 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Mild to Heavy Alcohol Consumption
Keywords: Pain; Elderly; Aged; Opioid; Cognition; Side-effects; Alcohol; Alcohol Use Disorder (AUD); Older
MeSH Terms: conditions — Pain; Alcoholism | interventions — Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, blood plasma, isolated DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Procedures: Study procedures include a screening visit, a study day visit, and a follow-up phone call. Oxycodone is administered on the study day.
  Interventions: Other: Oxycodone

INTERVENTIONS:
Other: Oxycodone — This study is interventional. Participants are given a single, one time administration of medication 10mg of oxycodone and observed

SUMMARY:
The purpose of this study is to examine the relationship between heavy alcohol use, pain, and response to pain medication in older adults.

DETAILED DESCRIPTION:
Potential participants complete a phone screen. If still found eligible, the participant comes in for 1 screening visit (3 hours long). Cognitive/problem solving tests, computerized tasks, CPT, questionnaires and functional measures are administered along with a screening blood lab. If a participant is eligible, he/she comes back for 1 full study day visit (9-10 hours long). A testing battery (similar to the one done during the screening visit) is completed at baseline and again at three timepoints following medication administration. Blood draws, vital signs, and pupil measurements are taken throughout the day. A follow-up phone call is completed within a few days of the full study day visit, during which a questionnaire is given.

ELIGIBILITY:
Inclusion Criteria:

* Age of 35 years old or above
* Mild to moderate pain
* alcohol consumption
* willingness to refrain from taking any sort of pain medication 24 hours prior to study visit as well as refraining from taking sedative-hypnotics, antihistamines, benzodiazepines, sleep aids, NSAIDs/opioid pain medications, alcohol, marijuana
* Cigarette smokers must be willing to refrain from smoking during the all day study visit

Exclusion Criteria:

* current regular use of an opioid or medications that involve the opioid receptor (naltrexone (vivitrol), buprenorphine (subutex), methadone (dolophine)
* abstains from alcohol
* unstable angina or CHF; cerebral vascular accident or recurrent TIAs in the prior 6 months, active cancer requiring current treatment, possible or probable dementia or mild cognitive impairment
* Diagnosis of schizophrenia or schizoaffective disorder, or anxiety disorder requiring regular medication
* History of recreational drug use in the past 1 year, excluding marijuana
* New or increased dose (within last 6 months) of CNS-active medications that may alter neurocognitive and/or psychomotor function: MAO inhibitors, neuroleptics, antidepressants, anticonvulsants, benzodiazepines, sleep aids
* Medications that may alter oxycodone metabolism: St. John's wort, Dilantin, tegretol, corticosteroids, rifampin
* Known hypersensitivity to oxycodone and other opioids;
* Pregnancy

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community dwelling participants in the greater Puget Sound region (Seattle and Tacoma) who consume alcohol on a frequent basis
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
response to a pain stimulus | given during study day
  Exposure to cold water, followed by exposure to warm water

SECONDARY OUTCOMES:
medication impact , opioid adjective checklist | Study day visit (9-10 hours long)
  adjective questionnaire on the impact of study medication scale of 0 t0 4 on likert scale
functional measure of balance modified berg balance test | Screening visit (3 hours long) and study day visit (9-10 hours long)
  score on a functional questionnaire (0 - 30)
Pupil size | Study day visit (9-10 hours long)
  measure of pupil diameter in millimeters
verbal memory performance on list learning task | Study day visit (9-10 hours long)
  immediate and delayed recall of a list of words (score of 0 - 45)

CONTACTS AND LOCATIONS:
Overall Officials: Monique M. Cherrier, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Univ. of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
For data obtained at UofW- a de-identified version can be made available upon request for data obtained at VAPSHCS IRB ISO, and PO do not allow the sharing of data, even de-identified data with other investigators- if VA regulations allow data sharing, then the investigators will be allowed to share data
Supporting Information: Study Protocol, SAP
Time Frame: upon completion of the study a copy of information will be made available on the open science framework site

REFERENCES:
- [Background] Cherrier MM, Amory JK, Ersek M, Risler L, Shen DD. Comparative cognitive and subjective side effects of immediate-release oxycodone in healthy middle-aged and older adults. J Pain. 2009 Oct;10(10):1038-50. doi: 10.1016/j.jpain.2009.03.017. Epub 2009 Sep 2. PMID 19729346

DOCUMENTS (1):
  • Informed Consent Form (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT02945293/ICF_000.pdf